CLINICAL TRIAL: NCT04727099
Title: Clinical Evaluation to Demonstrate the Safety and Performance of the Candela PicoWay System™
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Candela Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PWY20001
Record Dates: First submitted 2020-10-09; First posted 2021-01-27 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Wrinkle; Pigmented Lesions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Benign Pigmented Lesions (Experimental): Up to six (6) treatments with PicoWay laser for treatment of benign pigmented lesions
  Interventions: Device: PicoWay Laser System
- Wrinkles (Experimental): Up to six (6) treatments with PicoWay laser for treatment of wrinkles
  Interventions: Device: PicoWay Laser System

INTERVENTIONS:
Device: PicoWay Laser System — The PicoWay® laser system is an alexandrite laser pumped, solid-state Neodymium:Yttruium Aluminum Garnet (Nd:YAG) laser emitting energy at user selectable wavelengths of 1064 nm, 532 nm, 785 nm or 730 nm, designed for the treatment of tattoo, benign pigmented lesions, acne scars, and wrinkles.

SUMMARY:
This study is intended to demonstrate the safety and efficacy of the PicoWay™ Laser System for its intended uses: clearance of benign pigmented lesions and improvement in appearance of wrinkles.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, open-label study evaluating the safety and efficacy of the PicoWay™ Laser System for its intended uses: clearance of benign pigmented lesions and improvement in appearance of wrinkles.

Up to 200 eligible participants will be enrolled at up to five (5) sites. Participants will receive up to 6 treatments to the face and/or off-face locations with treatment intervals of 4 weeks +/- 2 weeks. Participants will complete follow-up visits for clinical evaluation and photography at 1 and 3 months after the final treatment. Total study duration is approximately 12 months (up to 9 months for treatment and 3 months for follow up).

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age or older
2. Willingness to provide signed, informed consent to participate in the study
3. Presence of mild or greater benign pigmented lesions, and/or wrinkles assessed as Fitzpatrick Wrinkle and Elastosis Score (FWS) >/= 1.
4. Willingness to adhere to study treatment and follow-up schedule
5. Willingness to adhere to post-treatment care instructions
6. Willingness to allow photographs and/or video of treated areas, and to release their use for scientific/educational and/or promotional/marketing purposes
7. Willing to abstain from any other procedures, medications or topicals in the study treatment areas for the duration of the study which the investigator deems would interfere with the study

Exclusion Criteria:

1. Pregnant, planning pregnancy during the study, or breast feeding
2. Tattooed skin in the intended treatment area unless tattoo removal treatment is to be performed.
3. Active sun tan in the intended treatment area
4. History of active Herpes Virus Simplex (HSV) or similar condition in the intended treatment area unless treated with prophylactic medication
5. History of melanoma
6. History of vitiligo in the intended treatment area
7. History of keloid or hypertrophic scar formation
8. History of Melasma in the intended treatment area per Investigator's discretion
9. Use of systemic retinoid therapy (e.g. Accutane) during the past 6 months
10. Severe immunosuppression resulting from medications and/or a medical condition that could impair healing after treatment
11. Open wound or infection in the intended treatment area
12. History of light induced seizure disorders
13. The subject is not suitable, in the opinion of the Investigator, for participation in the study due to inability to adhere to the study requirements, medical, or other reasons that could compromise the study integrity or subject safety
14. Dermatologic and/or cosmetic procedures including use of medications, or topicals in the intended treatment area(s) during a timepoint prior to the study that the investigator deems the subject unsuitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-09-28 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Benign Pigmented Lesions (BPLs) and Global Aesthetic Improvement Score (GAIS) | 12 months
  Improvement in Benign Pigmented Lesions (BPLs) from Baseline to 3 Month follow-up (= 12 months maximum) via the Investigator Global Aesthetic Improvement Score (IGAIS) where 5 = "worse," and 1 = "very much improved."
Benign Pigmented Lesions (BPLs) and Pigment Improvement Score (PIS) | 12 months
  Improvement in Benign Pigmented Lesions (BPLs) from Baseline to 3 Month follow-up (= 12 months maximum) via the Pigment Improvement Score (PIS) where a score of 0 = "no improvement" and a score of 4 = "Excellent response: Most or all lesions much lighter or gone"
Wrinkles and Global Aesthetic Improvement Score (GAIS) 3 month follow up | 12 months
  Improvement in the appearance of wrinkles from Baseline 3 Month follow-up (= 12 months maximum) via the Investigator Global Aesthetic Improvement Score (IGAIS) where 5 = "worse," and 1 = "very much improved."
Wrinkles and Fitzpatrick Wrinkle and Elastosis Score 3 month follow up | 12 months
  Improvement in the appearance of wrinkles from Baseline 3 Month follow-up (= 12 months maximum) via the Investigator Fitzpatrick Wrinkle and Elastosis Scale where a score of 1 = "fine wrinkles or mild elastosis" and 9 = "deep wrinkles or severe elastosis".

SECONDARY OUTCOMES:
BPLs and Global Aesthetic Improvement Score (GAIS) 1 month follow up | 10 months
  Improvement in BPLs from Baseline to 1 Month follow-up (= 10 months maximum) via the Investigator Global Aesthetic Improvement Score (IGAIS) where 5 = "worse," and 1 = "very much improved."
BPLs and PIS 3 month follow up | 10 months
  Improvement in BPLs from Baseline to 1 Month follow-up (= 10 months maximum) via the Pigment Improvement Score (PIS) where a score of 0 = "no improvement" and a score of 4 = "Excellent response: Most or all lesions much lighter or gone"
Wrinkles and Fitzpatrick Wrinkle and Elastosis Score 1 month follow up | 10 months
  Improvement in the appearance of wrinkles from Baseline to 1 Month follow-up (= 10 months maximum) via the Investigator Fitzpatrick Wrinkle and Elastosis Scale where a score of 1 = "fine wrinkles or mild elastosis" and 9 = "deep wrinkles or severe elastosis".
Wrinkles and Global Aesthetic Improvement Score (GAIS) 1 month follow up | 10 months
  Improvement in the appearance of wrinkles from Baseline to 1 Month follow-up (= 10 months maximum) via the Investigator Global Aesthetic Improvement Score (IGAIS) where 5 = "worse," and 1 = "very much improved."
Overall Subject Satisfaction 3 month follow up | 12 months
  Overall subject satisfaction with study treatments per treatment indication as measured by Subject Satisfaction Scale and Subject Global Aesthetic Improvement Score (SGAIS). (Baseline to 3 month follow up, approximately 12 months)

OTHER OUTCOMES:
Evaluation Adverse Events | through study completion, approximately 12 months
  Incidence, severity, and relatedness of adverse events. Severity is rated on a scale from 0 to 4 where 0 = none and 4 = severe

CONTACTS AND LOCATIONS:
Locations (1):
- Candela Institute of Excellence, Marlborough, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No IPD plan.